CLINICAL TRIAL: NCT05145049
Title: The Relationship of Anesthesia Method With Serum Lactate Level in Craniotomies
Status: Completed | Type: Observational
Sponsor: Ankara Diskapi Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Fatma Özkan Sipahioğlu, Principal Investigator, Anesthesiologist, Ankara Diskapi Training and Research Hospital
Other Study IDs: Lactate
Record Dates: First submitted 2021-11-08; First posted 2021-12-06 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Intracranial Neoplasm; Hyperlactatemia; Brain Tumor; Hypoperfusion
Keywords: hyperlactatemia; craniotomy; total intravenous anesthesia; general anesthesia
MeSH Terms: conditions — Brain Neoplasms; Hyperlactatemia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No

SUMMARY:
The investigators aimed to research the incidence of hyperlactatemia in craniotomy cases, the relationship of lactate elevation with tumor type and other factors that may be related, and whether the general anesthesia method applied (inhalation anesthesia or total ıntravenous anesthesia) affects lactate level.

DETAILED DESCRIPTION:
Lactate level is one of the easy-to-measure parameters that are frequently used in anesthesia and intensive care clinical practice, especially to evaluate the severity of disease and the response to treatment. In patients with high lactate levels, the first considerations are hypoperfusion and sepsis. However, many causes such as trauma, seizures, ischemia, diabetic ketoacidosis, thiamine deficiency, malignancies, liver dysfunction, genetic disorders, toxins, drugs, etc. can be associated with increased lactate. Many tissues in the body can produce lactate. 25% of production is from muscle, 25% skin, 20% brain, 20% RBC and 10% bowel cells. Some malignancies, especially hematological cancers, have also been associated with increased lactate. In recent years, it has been reported that serum lactate levels are associated with the degree of glial tumor malignancy, and that lactate can even be used as a non-invasive malignancy biomarker in brain tumors. In a recent study, it was reported that the type of 'glioblastoma multiforme' among patients who underwent craniotomy with the diagnosis of intracranial brain tumor was an independent influencer factor for preoperative and postoperative hyperlactatemia. Anesthesia is one of the factors that can affect lactate levels due to its effect on systemic perfusion and the hepatic effects of anesthetic drugs. It looks like that there is no study in the literature on the effect of anesthesia technique on hyperlactatemia in patients who underwent craniotomy. Therefore the investigators aimed to research the incidence of hyperlactatemia in craniotomy cases, the relationship of lactate elevation with tumor type and other factors that may be related, and whether the general anesthesia method applied (inhalation anesthesia or total ıntravenous anesthesia) affects lactate level.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled to undergo elective craniotomy for an intracranial mass
* adult patients

Exclusion Criteria:

* emergency
* In situations that may cause hyperlactatemia (such as sepsis, hepatic or renal failure, shock state, or patients who need inotropic support)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All patients who scheduled to undergo elective craniotomy for an intracranial mass older than 18 years old
Sampling Method: Probability Sample
Enrollment: 110 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2022-11-30 (Actual)

PRIMARY OUTCOMES:
lactate level | 0.hour
  basal lactate level via arterial blood gas at the beginning of surgery
lactate level | 1.hour
  lactate level via arterial blood gas at one hour after the beginning of surgery
lactate level | 3.hour
  lactate level via arterial blood gas at three hour after the beginning of surgery
lactate level | after extubation at the end of surgery
  lactate level via arterial blood gas at the end of the surgery

CONTACTS AND LOCATIONS:
Overall Officials: Fatma Özkan Sipahioglu, Principal Investigator — Ankara Diskapi Research and Training Hospital
Locations (1):
- Diskapi Training and Research Hospital, Ankara, Turkey (Türkiye)

REFERENCES:
- [Result] Andersen LW, Mackenhauer J, Roberts JC, Berg KM, Cocchi MN, Donnino MW. Etiology and therapeutic approach to elevated lactate levels. Mayo Clin Proc. 2013 Oct;88(10):1127-40. doi: 10.1016/j.mayocp.2013.06.012. PMID 24079682
- [Result] Branco M, Linhares P, Carvalho B, Santos P, Costa BM, Vaz R. Serum lactate levels are associated with glioma malignancy grade. Clin Neurol Neurosurg. 2019 Nov;186:105546. doi: 10.1016/j.clineuro.2019.105546. Epub 2019 Oct 1. PMID 31605893
- [Result] Bharadwaj S, Venkatraghavan L, Mariappan R, Ebinu J, Meng Y, Khan O, Tung T, Reyhani S, Bernstein M, Zadeh G. Serum lactate as a potential biomarker of non-glial brain tumors. J Clin Neurosci. 2015 Oct;22(10):1625-7. doi: 10.1016/j.jocn.2015.05.009. Epub 2015 Jun 19. PMID 26100160
- [Result] Mariappan R, Venkatraghavan L, Vertanian A, Agnihotri S, Cynthia S, Reyhani S, Tung T, Khan OH, Zadeh G. Serum lactate as a potential biomarker of malignancy in primary adult brain tumours. J Clin Neurosci. 2015 Jan;22(1):144-8. doi: 10.1016/j.jocn.2014.06.005. Epub 2014 Aug 27. PMID 25172017
- [Result] Ioannoni E, Grande G, Olivi A, Antonelli M, Caricato A, Montano N. Factors affecting serum lactate in patients with intracranial tumors - A report of our series and review of the literature. Surg Neurol Int. 2020 Mar 6;11:39. doi: 10.25259/SNI_552_2019. eCollection 2020. PMID 32257565